CLINICAL TRIAL: NCT01813357
Title: Does Rosuvastatin Delay Progression of Atherosclerosis in People With HIV Infection at Moderate Cardiovascular Risk? A Multicentre Randomized, Double Blind Placebo-controlled Trial
Brief Title: Does Rosuvastatin Delay Progression of Atherosclerosis in HIV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayside Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AH-491/12; ACTRN12612001082897 (Registry Identifier: Australian New Zealand clinical trials registry)
Record Dates: First submitted 2012-12-09; First posted 2013-03-19 (Estimated); Results first posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: HIV; Cardiovascular Disease
Keywords: HIV; Cardiovascular disease; Inflammation; Statin
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation | interventions — Rosuvastatin Calcium; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): sugar pill that is encapsulated so as to appear identical to the active agent
  Interventions: Other: Placebo
- Rosuvastatin (Experimental): Rosuvastatin 20mg daily
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — encapsulated tablet 20mg daily
  Other Names: Brand name: Crestor
  Arms: Rosuvastatin
Other: Placebo — Placebo arm included to maintain blinding
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
This study is a randomised double blind placebo controlled trial comparing Rosuvastatin with placebo in HIV positive people who are at intermediate cardiovascular risk.

It is possible that HIV positive people will receive a greater benefit from statins because of their higher baseline levels of inflammation. Current Australian guidelines recommend initiation of statin therapy on the basis of cholesterol level and the presence of other risk factors for heart disease (such as diabetes) but do not take into account whether a patient is infected with HIV. This study aims to determine what benefit HIV infected people will receive from starting statin therapy earlier then currently recommended.

DETAILED DESCRIPTION:
Participants will be randomised to receive either the active agent (Rosuvastatin) or a placebo once daily for 96 weeks.

Participants will undergo blood tests and ultrasounds of the arteries of the neck (carotid intima media thickness) prior to starting Rosuvastatin and then after 1 and 2 years on the drug to determine what effect it has on markers of inflammation, cholesterol levels and thickness of blood vessels.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Moderate cardiovascular disease (CVD) risk, (10-15% 10 year risk of CVD)
* HIV positive
* Stable combination anti-retroviral therapy (cART) with plasma HIV viral load <200copies/ml for ≥ 6 months

Exclusion Criteria:

* Recommended use of lipid lowering therapy according to Australian guidelines
* Prior use of statin, fibrate, ezetimibe within the last six months
* Contraindication to statin use

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2013-07-02 (Actual); Primary Completion 2018-05-17 (Actual); Study Completion 2018-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Hoy, Principal Investigator — Alfred health, Monash University
Locations (2):
- Alfred Hospital, Melbourne, Victoria, Australia
- Hospitaux Universitaires de Geneve, Geneva, Switzerland

REFERENCES:
- [Derived] Trevillyan JM, Dart A, Paul E, Cavassini M, Fehr J, Staehelin C, Dewar EM, Hoy JF, Calmy A. Impact of rosuvastatin on atherosclerosis in people with HIV at moderate cardiovascular risk: a randomised, controlled trial. AIDS. 2021 Mar 15;35(4):619-624. doi: 10.1097/QAD.0000000000002764. PMID 33252480

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Rosuvastatin
Started | 40 | 44
Completed | 35 | 38
Not Completed | 5 | 6
Not completed — Lost to Follow-up | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received daily placebo
- Active: Participants received daily rosuvastatin
- Total: Total of all reporting groups
Arm/Group | Placebo | Active | Total
Number analyzed (Participants) | 40 | 44 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (6.4) | 53.9 (5.9) | 54.1 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 40 | 42 | 82
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Australia | 27 | 28 | 55
  Switzerland | 13 | 16 | 29
Current Smoker [Count of Participants; unit: Participants] | 12 | 16 | 28
Total cholesterol [Mean (Standard Deviation); unit: mmol/L] | 5.3 (1.1) | 5.4 (0.8) | 5.3 (1.0)
Duration HIV infection [Mean (Standard Deviation); unit: years] | 13.6 (7.7) | 17.2 (8.5) | 16 (7.9)
Current cluster of differentiation of 4 (CD4) Cell count [Mean (Standard Deviation); unit: cells/ul] | 550 (254) | 693 (259) | 590 (250)

OUTCOME MEASURES:

1. Primary Outcome: Progression of Carotid Intima Media Thickness
Description: Carotid intima media thickness will be measured by ultrasonography and the change from baseline to week 96 calculated
Time Frame: Baseline to week 96
Population: Intention to treat
Measure: Mean (Standard Error); unit: mm
Arm/Group | Placebo | Rosuvastatin
Number analyzed (Participants) | 40 | 44
mm | 0.0062 (0.0039) | 0.004 (0.0036)
Statistical Analysis 1: Comparison: Placebo vs Rosuvastatin; Test type: Superiority; p = 0.684, Mixed Models Analysis; Mean Difference (Final Values) = 0.002

2. Secondary Outcome: Rates of Adverse Events
Description: Number of participants with adverse events in total and also the number of participants with adverse events thought secondary to the study medication
Time Frame: Will be assessed every 12 weeks and formally reported at 96 weeks of followup
Population: Intention to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rosuvastatin
Number analyzed (Participants) | 40 | 44
Participants | 22 | 35

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data was collected during study involvement and for 144 weeks post completion of last study visit (up to 240 weeks).
Description: Standard definitions used
Arm/Group | Placebo | Rosuvastatin
All-Cause Mortality (participants affected / at risk) | 0/40 | 1/44
Serious Adverse Events (participants affected / at risk) | 6/40 | 7/44
Other Adverse Events (participants affected / at risk) | 29/40 | 36/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=40) | Rosuvastatin (N=44)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
elevated creatinine kinase (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Type two diabetes (Endocrine disorders) | 0 (0) | 2 (2)
Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Elevated Alanine aminotransferase (ALT) (Hepatobiliary disorders) | 1 (1) | 1 (1) — Elevated ALT >5x Upper Limit of Normal
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Acute Mesentric Ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Oesophageal Malignancy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lumbar vertebral disc herniation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemoptysis (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=40) | Rosuvastatin (N=44)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 1 (1)
CK elevation (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
ALT elevation (Hepatobiliary disorders) | 4 (4) | 13 (13)
Non-specific gastrointestinal disturbance (Gastrointestinal disorders) | 4 (4) | 5 (5)
Hypertension (Cardiac disorders) | 11 (11) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2014-02-14): https://cdn.clinicaltrials.gov/large-docs/57/NCT01813357/Prot_SAP_ICF_000.pdf